CLINICAL TRIAL: NCT02305329
Title: Dosage Form Proportionality of Opicapone To-Be-Marketed Formulation in Healthy Subjects
Brief Title: Dosage Form Proportionality of Opicapone To-Be-Marketed Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-121
Record Dates: First submitted 2014-11-28; First posted 2014-12-02 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 BIA 9-1067 25 mg (Experimental): Period 1 - 5x5 mg OPC Period 2 - 1x25 mg OPC
  Interventions: Drug: BIA 9-1067
- Group 2 BIA 9-1067 25 mg (Experimental): Period 1 - 1x25 mg OPC Period 2 - 5x5 mg OPC
  Interventions: Drug: BIA 9-1067
- Group 1 BIA 9-1067 50 mg (Experimental): Period 1 - 2x25 mg OPC Period 2 - 1x50 mg OPC
  Interventions: Drug: BIA 9-1067
- Group 2 BIA 9-1067 50 mg (Experimental): Period 1 - 1x50 mg OPC Period 2 - 2x25 mg OPC
  Interventions: Drug: BIA 9-1067

INTERVENTIONS:
Drug: BIA 9-1067
  Other Names: OPC, Opicapone

SUMMARY:
Single-centre, open-label, randomized, two-sequence, two-way crossover study. The study consisted of two consecutive single-dose treatment periods separated by a washout period of 10 to 14 days or more.

DETAILED DESCRIPTION:
Single-centre, open-label, randomized, two-sequence, two-way crossover study. The study consisted of two consecutive single-dose treatment periods separated by a washout period of 10 to 14 days or more. In Group 1 the volunteers received a single oral dose of 25 mg OPC. In Group 2 the volunteers received a single oral dose of 50 mg OPC

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 45 years, inclusive;
* Body mass index (BMI) between 19 and 30 kg/m²;
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination, and 12-lead ECG; - Negative tests for hepatitis B surface antigen (HBsAg), anti-hepatitis C vírus (anti-HCV) antibodies, and anti-human immunodeficiency virus (HIV)-1/-2 antibodies at screening;
* Clinical laboratory test results clinically acceptable at screening and admission to each treatment period;
* Negative screen for alcohol and drugs of abuse at screening and admission to each treatment period;
* Non-smokers or ex-smokers for at least 3 months;
* Able and willing to give written informed consent;
* If female: She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used an effective nonhormonal method of contraception (intrauterine device or intrauterine system; condom or occlusive cap [diaphragm or cervical or vault caps] with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomized male partner, provided that he was the sole partner of that subject) for all the duration of the study; and she had a negative serum pregnancy test at screening and a negative urine pregnancy test on Day -1 of each treatment period.

Exclusion Criteria:

* A clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders;
* A clinically relevant surgical history;
* Any clinically relevant abnormality in the coagulation tests;
* Any clinically relevant abnormality in the liver function tests. If the subject had a borderline clinically relevant abnormality that was not considered clinically significant, a retest could be done after discussion with the sponsor's medical monitor;
* A history of relevant atopy or drug hypersensitivity;
* A history of alcoholism or drug abuse;
* Consume more than 14 units of alcohol a week;
* A significant infection or known inflammatory process on screening or admission to each treatment period;
* Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period;
* Used medicines within 2 weeks of admission to first period that could have affected the subject's safety or other study assessments in the investigator's opinion;
* Previously received OPC. Previous use of OPC was documented by questioning the subjects;
* Used any investigational drug or participated in any clinical trial within 90 days prior to screening
* Participated in more than 2 clinical trials within the 12 months prior to screening;
* Donated or received any blood or blood products within the 3 months prior to screening;
* Vegetarians, vegans or have medical dietary restrictions;
* Not able to communicate reliably with the investigator;
* Unlikely to co-operate with the requirements of the study; unwilling or unable to give written informed consent;
* If female: she was pregnant or breast-feeding; she had a positive serum pregnancy test; she was of childbearing potential and did not use an accepted effective contraceptive method or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 BIA 9-1067 25 mg: Period 1 - 5x5 mg OPC Period 2 - 1x25 mg OPC
  BIA 9-1067
- Group 2 BIA 9-1067 25 mg: Period 1 - 1x25 mg OPC Period 2 - 5x5 mg OPC
  BIA 9-1067
- Group 1 BIA 9-1067 50 mg: Period 1 - 2x25 mg OPC Period 2 - 1x50 mg OPC
  BIA 9-1067
- Group 2 BIA 9-1067 50 mg: Period 1 - 1x50 mg OPC Period 2 - 2x25 mg OPC
  BIA 9-1067
Period: Overall Study
Arm/Group | Group 1 BIA 9-1067 25 mg | Group 2 BIA 9-1067 25 mg | Group 1 BIA 9-1067 50 mg | Group 2 BIA 9-1067 50 mg
Started | 14 | 14 | 14 | 14
Period 1 | 14 | 14 | 14 | 14
Period 2 | 14 | 13 | 14 | 14
Completed | 14 | 13 | 14 | 14
Not Completed | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 BIA 9-1067 25 mg | Group 2 BIA 9-1067 25 mg | Group 1 BIA 9-1067 50 mg | Group 2 BIA 9-1067 50 mg | Total
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 14 | 14 | 56
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 7 | 7 | 28
  Male | 7 | 7 | 7 | 7 | 28

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration of 9-1067
Description: Cmax - maximum observed plasma concentration of 9-1067.
Time Frame: before OPC dosing, and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48h post-OPC dose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 5x5mg BIA 9-1067: 5x5mg BIA 9-1067, OPC
- 1x25 mg BIA 9-1067: 1x25 mg BIA 9-1067, OPC
- 2x25 mg BIA 9-1067: 2x25 mg BIA 9-1067, OPC
- 1x50 mg BIA 9-1067: 1x50 mg BIA 9-1067, OPC
Arm/Group | 5x5mg BIA 9-1067 | 1x25 mg BIA 9-1067 | 2x25 mg BIA 9-1067 | 1x50 mg BIA 9-1067
Number analyzed (Participants) | 27 | 28 | 28 | 28
ng/mL | 600 (221) | 567 (222) | 955 (297) | 917 (426)

2. Secondary Outcome: Tmax - Time of Occurrence of Cmax of 9-1067
Description: tmax - time of occurrence of Maximum Observed Plasma Concentration of 9-1067
Time Frame: before OPC dosing, and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48h post-OPC dose
Measure: Median (Full Range); unit: hours
Arm/Group | 5x5mg BIA 9-1067 | 1x25 mg BIA 9-1067 | 2x25 mg BIA 9-1067 | 1x50 mg BIA 9-1067
Number analyzed (Participants) | 27 | 28 | 28 | 28
hours | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00] | 2.00 [0.50 to 8.00]

3. Secondary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve Calculated Between Time of Administration and Time t
Time Frame: before OPC dosing, and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48h post-OPC dose
Measure: Mean (Standard Deviation); unit: h.ng/mL
Arm/Group | 5x5mg BIA 9-1067 | 1x25 mg BIA 9-1067 | 2x25 mg BIA 9-1067 | 1x50 mg BIA 9-1067
Number analyzed (Participants) | 27 | 28 | 28 | 28
h.ng/mL | 1603 (566) | 1461 (529) | 2669 (945) | 2539 (1066)

4. Secondary Outcome: AUC0-∞ - Area Under the Plasma Concentration-time Curve Extrapolated to Infinity
Description: AUC0-∞ - Area under the plasma concentration-time curve extrapolated to infinity.
Time Frame: before OPC dosing, and 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36 and 48h post-OPC dose
Measure: Mean (Standard Deviation); unit: h.ng/mL
Arm/Group | 5x5mg BIA 9-1067 | 1x25 mg BIA 9-1067 | 2x25 mg BIA 9-1067 | 1x50 mg BIA 9-1067
Number analyzed (Participants) | 27 | 28 | 28 | 28
h.ng/mL | 1679 (586) | 1539 (554) | 2699 (1012) | 2612 (1082)

ADVERSE EVENTS:
Arm/Group | 5x5mg BIA 9-1067 | 1x25 mg BIA 9-1067 | 2x25 mg BIA 9-1067 | 1x50 mg BIA 9-1067
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 7/27 | 11/28 | 12/28 | 15/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5x5mg BIA 9-1067 (N=27) | 1x25 mg BIA 9-1067 (N=28) | 2x25 mg BIA 9-1067 (N=28) | 1x50 mg BIA 9-1067 (N=28)
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 1
Influenza like illness (General disorders) | 2 | 1 | 1 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 3
Headache (Nervous system disorders) | 3 | 5 | 6 | 4
Somnolence (Nervous system disorders) | 0 | 2 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 1 | 1
VOMITING (Gastrointestinal disorders) | 1 | 0 | 1 | 1
CATHETER SITE PAIN (General disorders) | 0 | 0 | 0 | 1
BACTERIAL VAGINOSIS (Infections and infestations) | 0 | 0 | 0 | 1
ORAL HERPES (Infections and infestations) | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 0 | 1
TENSION HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 1
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other